CLINICAL TRIAL: NCT03579901
Title: Study of the Safety and Effectiveness of the Motiva Implants® Silicone Gel-Filled Breast Implants SmoothSilk® in Subjects Who Are Undergoing Primary Breast Augmentation, Primary Breast Reconstruction, and Revision Surgery
Brief Title: Study of the Safety and Effectiveness of Motiva Implants®
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Motiva USA LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLIN-17-008
Record Dates: First submitted 2018-04-12; First posted 2018-07-09 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Breast Implants
Keywords: Breast Implants; Breast Surgery; Breast Augmentation; Breast Reconstruction

STUDY DESIGN:
Intervention Model Description: Multicenter Single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Primary Breast Augmentation (Other): Subjects age 22 and over, indicated to increase breast size
  Interventions: Device: Silicone gel-filled breast implants - Motiva Implants® Investigational breast implants
- Primary Breast Reconstruction (Other): Subjects age 18 and over, Surgery to replace breast tissue that has been removed due to cancer, prophylactic mastectomy, breast trauma or that has failed to develop properly due to a severe breast anomaly.
  Interventions: Device: Silicone gel-filled breast implants - Motiva Implants® Investigational breast implants
- Revision Augmentation (Other): Revision surgery to correct or improve the results of a previous breast augmentation
  Interventions: Device: Silicone gel-filled breast implants - Motiva Implants® Investigational breast implants
- Revision Reconstruction (Other): Revision surgery to correct or improve the results of a previous breast reconstruction.
  Interventions: Device: Silicone gel-filled breast implants - Motiva Implants® Investigational breast implants

INTERVENTIONS:
Device: Silicone gel-filled breast implants - Motiva Implants® Investigational breast implants — Breast augmentation

SUMMARY:
This study evaluates the safety and effectiveness Motiva Implants® in women who are undergoing primary breast augmentation, primary breast reconstruction or revision breast surgery.

DETAILED DESCRIPTION:
Prospective, Single Arm, Multicenter Study. Following FDA approval, follow-up data will continue to be collected for all cohorts on adverse events, reoperations, patient satisfaction, physician satisfaction and quality of life for a total of 10 years.

ELIGIBILITY:
Inclusion Criteria

* Genetic female.
* Patient is seeking one of the following procedures:

Primary Breast Augmentation Primary Breast Reconstruction Revision Augmentation Revision Reconstruction

* Patient has adequate tissue available to cover implant(s).
* Willingness to follow all study requirements including agreeing to attend all required follow-up visits and signs the informed consent.
* Agrees to have device returned to Establishment Labs if explanted.
* Willing to undergo Magnetic Resonance Imaging (MRI) evaluation of medically advised.

Exclusion Criteria:

* Has any breast disease considered to be pre-malignant in one or both breasts or is reporting mutations in BRCA1 or BRCA2 without a previous bilateral mastectomy or an untreated cancer of any type.
* Has inadequate or unsuitable tissue (e.g., due to radiation damage, ulceration compromised vascularity, history of compromised wound healing).
* Has an abscess or infection.
* Is pregnant or nursing or has had a full-term pregnancy or lactated within 6 months of enrollment.
* Is taking any drugs that would interfere with blood clotting, or that might result in elevated risk and or significant postoperative complications.
* Has any medical condition such as obesity (BMI ≥ 40), diabetes, autoimmune disease, chronic lung or severe cardiovascular disease that might result in unduly high surgical risk and or significant postoperative complications.
* Has any connective tissue/autoimmune disorder or rheumatoid disease, such as systemic lupus erythematosus, discoid lupus, scleroderma, or rheumatoid arthritis, among others.
* Has any condition that impedes the use of magnetic resonance imaging (MRI) including implanted metal device, claustrophobia or other conditions that would make MRI scan prohibited.
* Has a history of psychological characteristics that are unrealistic or unreasonable given the risks involved with the surgical procedure.
* Has been implanted with any non-FDA approved breast implant.
* Has been implanted with any silicone implant other than breast implants.
* HIV positive (based on medical history).
* Has been diagnosed with anaplastic large cell lymphoma (ALCL).
* Works for Establishment Labs, Motiva USA or any of their subsidiaries, the study surgeon, or ICON the Contract Research Organization (CRO) that is helping to conduct the study or are directly-related to anyone that works for Establishment Labs, Motiva USA or any of their subsidiaries, the study surgeon, or the CRO.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 800 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2032-08-30 (Estimated); Study Completion 2033-02-28 (Estimated)

PRIMARY OUTCOMES:
Analyze and report the total adverse events rate ("any complication)" of the Silicone Gel filled Motiva Implants®. Kaplan-Meier analysis of adverse events will be conducted by time period for each type of adverse event. | 10 Years
Analyze patient satisfaction on a 5-point Likert scale post-implant for all implantation groups. | 10 Years

SECONDARY OUTCOMES:
Kaplan-Meier analysis of all complications, including reoperation and explantation | 10 Years
Cox regression analyses for the following endpoints: Capsular contracture III/IV, Breast Pain, Infection, and Implant Rupture | 10 Years
Kaplan-Meier analysis of rupture. | 10 Years
Kaplan-Meier analysis of connective tissue disease (CTD) and CTD signs/symptoms | 10 Years
Kaplan-Meier analysis of Cancer (Breast Cancer, Breast Implant-Associated Anaplastic Large Cell Lymphoma (BIA-ALCL), and others) | 10 Years
Patient Satisfaction with Breast (BREAST-Q™) Questionnaire | 10 Years
Physician Satisfaction (5-point Likert scale) | 10 Years
Validated Quality of Life questionnaires | 10 Years
Breast Measurements (Net Chest Circumference and Hemi-Circumference) change from baseline | 10 Years

CONTACTS AND LOCATIONS:
Locations (29):
- United States (27):
  - Gerald Minitti, MD, FACS, Beverly Hills, California
  - Steven Teitelbaum, MD, FACS, Santa Monica, California
  - Westlake Cosmetic Surgery Center, Westlake Village, California
  - The Center for Cosmetic Surgery, Golden, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Plastic Surgery, Chicago, Illinois
  - Northwestern Specialists in Plastic Surgery, S.C., Chicago, Illinois
  - Meridian Plastic Surgery Center, Indianapolis, Indiana
  - CaloAesthetics® Plastic Surgery Center, Louisville, Kentucky
  - The Wall Center for Plastic Surgery, Shreveport, Louisiana
  - Partners in Plastic Surgery of West Michigan, Grand Rapids, Michigan
  - Parkcrest Plastic Surgery, St Louis, Missouri
  - Glicksman Plastic Surgery, Sea Girt, New Jersey
  - Mark D. Epstein, MD, FACS/ Center for Aesthetic Surgery, Hauppauge, New York
  - NYU Plastic Surgery Associates, New York, New York
  - May Center for Mount Sinai Doctors, New York, New York
  - Fifth Avenue Millennium Aesthetic Surgery, PLLC, New York, New York
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Movassaghi Plastic Surgery & Ziba Medical Spa, Eugene, Oregon
  - Portland Plastic Surgery, Portland, Oregon
  - Body by Z, Providence, Rhode Island
  - Maxwell Aesthetics, PLLC, Nashville, Tennessee
  - Strock Plastic Surgery, Fort Worth, Texas
  - Houston Methodist, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - William P. Adams Plastic Surgery, University Park, Texas
  - PeaceHealth Plastic Surgery, Vancouver, Washington
- Plastische Chirurgie im Medienhafen, Düsseldorf, Germany
- Victoriakliniken, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No